CLINICAL TRIAL: NCT05151809
Title: Multicenter, Nationwide, Observational, Retrospective and Prospective Study Based on the Development of a Patients Database Linked to a Biological Sample Storage
Brief Title: National Database on Primary Biliary Cholangitis
Acronym: PBC322
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: PBC322
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis; Disease phenotypes; National Database
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Clinical Laboratory Information Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Biological samples are collected at time of recruitment and on a yearly basis (for blood, urine and stools).The collection of bile and liver tissue depends on the specific procedures (ERCP and liver biopsy) that are performed based on clinical needs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PBC population residing in Italy: All PBC patients living in Italy and aged at least 18 years can be included in the database. According to well-established criteria, PBC is diagnosed in subjects who fulfill two of the three of following criteria:
  1. elevated alkaline phosphatase and /or GGT;
  2. positive anti-mitochondrial autoantibodies (titer ≥ 1:40) or PBC-specific antinuclear antibodies (gp-210 and sp100);
  3. characteristic histological features of florid bile ducts lesions and granulomatous lesion.
  Interventions: Other: Clinical information

INTERVENTIONS:
Other: Clinical information — The investigators will recruit PBC patients and collect important clinical information and laboratory investigation, together with biological samples.
  Other Names: Laboratory information; Biological samples

SUMMARY:
Primary biliary cholangitis (PBC) is a rare, autoimmune, cholestatic liver disease. No data about the disease epidemiology exist in Italy. Therefore this study aims to develop a national PBC patient database linked to a biological sample storage.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC) is an immune-mediated liver disease characterized by chronic inflammation of the intrahepatic bile ducts, causing progressive ductopenia, cholestasis, and if not effectively treated, leading to fibrosis, cirrhosis and liver failure. Nowadays almost all patients with PBC are diagnosed at an early disease stage and receive treatment with ursodeoxycholic acid (UDCA) which is currently the only drug approved for the treatment of patients with PBC. However, approximately 20% to 30% (up to >50% in patients presenting under the age of 40 years) still does not have a benefit from UDCA and has a reduced prognosis as compared to healthy individuals. Major steps forwards in the field of PBC have been done in the last decade, however there are still significant areas of unmet clinical need in PBC: the lack of knowledge on etiopathogenesis; a poor understanding of disease sub-phenotypes; the lack of biomarkers of disease progression that allow risk stratification needed in clinical management and trials design, among the others. In the current evolving research landscape with the availability of the -omics technologies generating libraries of genome-wide data, metabolomics and proteomics data, among the others, the prospects of discovering the gene and molecular underpinnings of PBC are more promising than ever. Scientists envision an era of "personalized medicine" when more and more people will obtain their own genetic and metabolic maps, enabling them to identify their status as carriers of specific risk profiles.

Based on these premises, the current project aims to build up a research, nation-wide infrastructure (around 60 Italian participating centres will be involved) to study the biology of PBC and, in particular, to explore why a significant group of, typically young patients fail primary therapy with UDCA, placing them at risk of developing progressive disease and needing liver transplantation (LT). The investigators will recruit patients and organise the collection of important clinical information and laboratory investigation, together with biological samples. Data will be collected in the form of electronic Case Report Forms (REDCap cloud) that will be completed by clinicians at baseline and thereafter on an annual basis. The clinical information will allow us to identify patients' clinical profiles. The biological samples will allow to understand key aspects of people's make up, including patient genes and the way their immune system works, and the differences in make up between people with different clinical phenotypes.

This research infrastructure would represent an invaluable resource for successful translational research in this field. Specifically, it would serve investigators conducting research; clinicians treating patients; epidemiologists gathering demographic data; and the drug and device industry seeking new markets. It also can represent a necessary infrastructure for the implementation of the European Reference Networks (ERN) for rare diseases, main pillars of the current EU policy framework on National Plans for research and development. The Italian PBC database would also be crucial for drug development, specifically to assess the feasibility of clinical trials, to facilitate the planning of appropriate clinical trials, to support the enrolment of patients and to assess the impact of new interventions.

ELIGIBILITY:
Inclusion Criteria:

All PBC patients living in Italy and aged at least 18 years can be included in the database. According to well-established criteria, PBC is diagnosed in subjects who fulfill two of the three of following criteria:

* elevated alkaline phosphatase and /or GGT;
* positive anti-mitochondrial autoantibodies (titer ≥ 1:40) or PBC-specific antinuclear antibodies (gp-210 and sp100);
* characteristic histological features of florid bile ducts lesions and granulomatous lesion.

Exclusion Criteria:

The patient has explicitly declared his/her unwillingness to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the italian patients fulfilling the diagnostic criteria for Primary Biliary Cholangitis (European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67) and aged at least 18.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2029-01-24 (Estimated); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Phenotypes and sub-phenotypes of PBC Italian patients | Overall duration of the study (10 years)
  Identify and define distinct phenotypes and sub-phenotypes of PBC patients at higher risk of disease progression.

SECONDARY OUTCOMES:
Response to UDCA therapy | Overall duration of the study (10 years)
  Defined as Alkaline Phosphatase Level<1 x upper limit of normal. The investigators will fit a multivariate analysis using logistic regression using baseline variables.
Identification of factors influencing the progression of PBC | Overall duration of the study (10 years)
  The investigators will calculate the time from the diagnosis of PBC to an event (liver decompensation, liver transplantation or death). They will then fit a multivariate analysis using Cox's proportional hazards regression model of diverse explanatory variables available at baseline.
Safety and long-term efficacy of novel therapies | Overall duration of the study (10 years)
  The investigators will evaluate prospectively laboratory investigation and the treatment response to novel therapies that are entering the clinical practice, e.g. obeticholic acid, fibrates.

CONTACTS AND LOCATIONS:
Locations (55):
- Italy (55):
  - Ospedali riuniti di Ancona, Ancona
  - A.O.U. Consorziale - Policlinico Bari- UO Gastroenterologia, Bari
  - UO di gastroenterologia, Asst Papa Giovanni XXIII, Bergamo
  - Policlinico S. Orsola Malpighi- UO Medicina Interna, Bologna
  - Policlinico S.Orsola Malpighi- Ambulatorio di epatologia e gestione trapianto epatico, Bologna
  - Gastroenterologia, fisiopatologia e endoscopia digestiva, Azienda sanitaria dell'alto adige, Bolzano
  - Unità epatologica ed ecografia internistica a valenza dipartimentale, Fondazione Ospedaliera Poliambulanza, Brescia
  - UO di gastroenterologia, Spedali civili di Brescia, Brescia
  - UO epatologia, Azienda ospedaliero università di Cagliari Policlinico universitario Monserrato, Cagliari
  - Ospedale IRCCS Saverio De Bellis- UOC di Gastroenterologia 1, Castellana Grotte
  - UO epatologia Ospedale Garibaldi, Catania
  - UO di fisiopatologia digestiva, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
  - UO di gastroenterologia, Ospedale Valduce, Como
  - Azienda Socio Sanitaria Territoriale (ASST) di Cremona- UO Medicina Interna - Ambulatori di Epatologia, Cremona
  - Presidio Ospedaliero di Faenza- UO Medicina Interna, Faenza
  - UO Clinica Medica, Azienda Ospedaliera Universitaria Careggi Firenze, Florence
  - Centro C.U.R.E. Centro Universitario per la ricerca e la Cura delle Malattie Epatiche, Foggia
  - Ambulatorio di Malattie del Fegato, U.O. Medicina, ASST Valle Olona, Presidio di Gallarate, Gallarate
  - UO Clinica Gastroenterologica, Policlinico San Martino, Genova
  - Centro Medicina del Viaggiatore e delle Migrazioni, ASP Catanzaro, Presìdio Ospedaliero "Giovanni Paolo II", Lamezia Terme
  - UO di epatologia clinica e biomolecolare, Università degli studi di Messina, Messina
  - University of Milano-Bicocca, Milan
  - Policlinico di Milano, Milan
  - UO di epatologia, Ospedale Niguarda Ca' Granda, Milan
  - UO di Epatologia, Ospedale San Giuseppe, Milan
  - UO epatologia, Istituto scientifico universitario San Raffaele, Milan
  - AOU di Modena- U.O. Gastroenterologia, Modena
  - Struttura Complessa di Medicina ad Indirizzo Metabolico Nutrizionale, Dipartimento Ospedaliero di Medicina Interna, Modena
  - Day Hospital e Ambulatorio di Epatoogia e Nutrizione Clinica, Fondazione Evangelica Villa Betania, Ospedale generale di Zona, Napoli
  - Ospedale policlinico Federico II di Napoli, Napoli
  - Università della Campania Luigi Vanvitelli di Napoli- Dipartimento di epato-gastroenterologia, Napoli
  - UO medicina ed epatologia, Ospedale maggiore della carità, Novara
  - UO di Gastroenterologia, Azienda ospedaliera di Padova, Padua
  - UO di Medicina Interna, Azienda Ospedaliera di Padova, Padua
  - UO gastroenterologia, Policlinico Paolo Giaccone, Palermo
  - Malattie infettive ed epatologia, Azienda ospedaliero universitaria di Parma, Parma
  - Day Hospital Internistico e ambulatorio di Epatologia, ASL Pescara, Pescara
  - UO epatologia, AOU pisana Cisanello, Pisa
  - S.C. Gastroenterologia, Ospedale di Pordenone, AS FO, Pordenone
  - Medicina clinica ed epatologia, Policlinico universitario campus bio-medico, Roma
  - Policlinico Universitario Fondazione Agostino Gemelli- UO di medicina interna, Roma
  - UO di Epatologia, Universita' di Roma Tor Vergata, Roma
  - UO di Gastroenterologia, Policlinico Umberto I, Roma
  - Medicina interna ed epatologia, Istituto clinico Humanitas, Rozzano
  - Università degli studi di Salerno, Salerno
  - SSD Epatologia, Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - UO di Gastroenterologia e Endoscopia Digestiva, Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedale Universitaria di Sassari- UOC Medicina Interna, Sassari
  - S.C. Gastroenterologia, Azienda Ospedaliero-Universitaria Molinette, Torino
  - Gastroenterologia ed endoscopia digestiva, Azienda provinciale per i servizi sanitari, Trento
  - Ospedale regionale Ca' Foncello di Treviso- Unità operativa complessa di Gastroenterologia, Treviso
  - SC (UCO) Clinica Patologie del Fegato, Ospedale di Cattinara, ASU GI, Trieste
  - SOS di DPT Epatologia e Trapianti di Fegato, ASU FC, Udine
  - UO di gastroenterologia ed endoscopia digestiva, Azienda macchi, Asst sette laghi, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona- UOC Gastroeneterologia A, Verona

IPD SHARING:
Plan to Share IPD: No